CLINICAL TRIAL: NCT01171911
Title: Nanjing First Hospital, Nanjing Medical University
Brief Title: Comparison of Intravenous Injection of Calcium Antagonist and Beta-blockade on Endothelial Shear Stress of Coronary Artery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Shao-Liang Chen/Hospital director, Nanjing First Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NJESS20103079
Record Dates: First submitted 2010-07-23; First posted 2010-07-29 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2010-04

CONDITIONS: Acute Coronary Syndrome; Coronary Artery Disease
Keywords: Endothelial shear stress; Calcium channel blocker
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease | interventions — Nicardipine; esmolol; Calcium Channel Blockers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Nicardipine , Esmolol — A loading dose of Nicardipine 10mg was at a bolus injected through vein , then continuous trans-venous titration at a speed 1ug/kg was kept. A loading dose of Esmolol 0.5mg/kg/min was at a bolus injected through vein , then continuous trans-venous titration at a speed 0.2mg/kg/min was kept.
  Other Names: Calcium channel blocker

SUMMARY:
Both calcium channel antagonist and beta-blocker have cardioprotective effect. Endothelial shear stress is predictive factor of clinical outcomes in patients with obstructive stenosis.

The present study aims at comparing the re-distribution of shear stress and blood velocity during whole cardiac cycle after trans-coronary injection of Nicardipine and esmolol.

DETAILED DESCRIPTION:
Blood flow-induced endothelial shear stress has strong effect on endothelial function and development or progression of plaque formation. It is extensively accepted that low and/or oscillating shear stress causes endothelial dysfunction and is one of crucial factors in localizing early atherosclerosis .In contrary, normal and high shear stress is atheroma protective and is involved in compensatory remodeling . Most studies reported that the endothelial shear stress distribution in often idealized geometrical models of human coronary arteries was the subject of numerous investigations , and in these studies it was shown that the geometry of coronary arteries is the main determinant of the observed shear stress distribution. Generally, downstream of a plaque, low shear stress can be expected, Several cardiovascular active drugs have been shown to be cardio-protective for patients with obstructive coronary disease. Of these drugs, calcium channel blocker is one of most prescribed in everyday clinical practice. Ninomiya et al. reported calcium channel blocker was associated with increased coronary diameter and blood fluid with dose-dependent pattern in patients with normal or mild stenotic coronary artery. However, no reports on the dynamic change of endothelial shear stress after calcium channel blocker in -vitron were published so far. As a result, the aim of this study was to evaluate the effect of intra-venous injection of Nicardipine, one calcium channel blocker with shorter half-time, on the re-distribution of endothelial shear stress in patients with acute coronary syndrome and mild stenotic (<50%) coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unstable angina and non-Q wave myocardial infarction
* Age 18-75 yr.
* Diameter stenosis of coronary artery<70% diameter stenosis by visual estimation
* Blood pressure >110/70 mmHg
* Heart rate 60-~100 bpm, No cardiac arrhythmias

Exclusion Criteria:

* St-elevation myocardial infarction
* Lower blood pressure(<100/70mmHg)
* Heart rate <60 or >100 bpm, The presence of cardiac arrhythmias
* Allergy to study drugs
* Women in pregnancy
* Liver dysfunction
* Creatinine >2.5mg/dl
* Bleeding stroke within 6 months
* Left ventricular ejection fraction<30% before maximal medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Endothelial shear stress assessed by computational fluid dynamics | After four minutes
  At the peak effect of drug that the mean blood pressure (MBP) reduced by 10% or more, or the heart rate increased by 10-15 bpm.

SECONDARY OUTCOMES:
Minimal lumen area by intravascular ultrasound | After four minutes
  At the peak effect of drug that the mean blood pressure (MBP) reduced by 10% or more, or the heart rate increased by 10-15 bpm.

CONTACTS AND LOCATIONS:
Overall Officials: Shao-liang Chen, Director, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital,Nanjing Medical University, Nanjing, Jiangsu, China